CLINICAL TRIAL: NCT01902433
Title: Astym® Treatment Compared With Eccentric Exercise in the Management of Chronic Mid-substance Achilles Tendinopathy: A Multisite a Randomized Controlled Trial
Brief Title: Astym® Compared Eccentric Exercise for Chronic Mid-substance Achilles Tendinopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We were unable to recruit participants to the study
Sponsor: Emily Slaven, PT, PhD (Other)
Collaborators: Performance Dynamics (Unknown)
Responsible Party: Sponsor-Investigator, Emily Slaven, PT, PhD, Assistant Professor, University of Indianapolis
Organization: University of Indianapolis (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASTYM2013
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Achilles Tendon Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Astym (Experimental): A form of soft tissue mobilization using instruments
  Interventions: Procedure: Astym
- Eccentric Exercise (Active Comparator): Eccentric exercise is a form of exercise where the benefit comes from applying a controlled lengthening stress to the muscle and tendon.
  Interventions: Procedure: Astym

INTERVENTIONS:
Procedure: Astym

SUMMARY:
The purpose of this study is to compare the changes in pain and self-perceived function between two different treatments for Achilles tendinopathy: the Astym® protocol (a form of soft tissue mobilization using instruments) and a specific exercise protocol that involves strengthening the calf and Achilles tendon. Astym® (A-stim) is not an acronym, but rather stands for "A Stimulation" of the body's healing response, describing the physiologic process which occurs with Astym treatment. Astym is the trademark name of a non-invasive treatment where instruments are applied topically to locate unhealthy soft tissue, and to transfer mild to moderate pressure to the underlying soft tissue structures. The aim of Astym treatment is to eliminate scar tissue and stimulate tissue regeneration. Both the principal investigator and co-investigator have been trained and certified in administering the Astym treatment. The specific exercise protocol will involve exercises that strengthen the Achilles and calf through eccentric exercise. Eccentric exercise is a form of exercise where the benefit comes from applying a controlled lengthening stress to the muscle and tendon.

ELIGIBILITY:
Inclusion Criteria

* Pain for 3 months or longer in the mid portion of only one Achilles tendon.
* Must read, speak and understand English

Exclusion Criteria

* Previous surgery to the Achilles tendon that is currently painful
* An injection into the Achilles tendon in the previous 4 weeks
* Have symptoms in both Achilles tendons concurrently
* Have taken fluoroquinolone antibiotics in the past 6 months

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
VISA-A | 1 year

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Slaven, PhD, Principal Investigator — University of Indianapolis
Locations (2):
- United States (2):
  - IU Health, Indianapolis, Indiana
  - Utah Physical Therapy, Lehi, Utah

IPD SHARING:
Plan to Share IPD: Undecided
Only two participants were recruited to the study at the closure of the study